CLINICAL TRIAL: NCT00875108
Title: An Open Label, Multi-Center, Follow-on Study Examining the Long-Term Safety and Efficacy of Insulin VIAject™ in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIAject™-09J
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIAject™ (Experimental): Single injection
  Interventions: Drug: VIAject™

INTERVENTIONS:
Drug: VIAject™ — Subcutaneous injection 25 IU/mL

SUMMARY:
Follow-on study to the VIAject™-08J study to evaluate the long-term safety and efficacy of VIAject™ when used as prandial insulin in combination with Lantus® in subjects with type 2 diabetes mellitus.

The VIAject™-08J study is the efficacy and safety study for insulin VIAject™ to demonstrate equivalent blood glucose control in patients with type 2 diabetes mellitus with VIAject™ insulin or regular human insulin as prandial insulin and to demonstrate an equivalent safety profile for VIAject™ in comparison to human insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the VIAject™-08J protocol
2. Informed consent must be obtained in writing for all subjects.

Exclusion Criteria:

1. History of frequent severe hypoglycemia within the prior six months which prevent study participation at the discretion of the investigator
2. History of known hypersensitivity to any of the components in the study medication
3. Progressive disease likely to prove fatal
4. Known significant hepatic disease or serum AST or ALT values > 3 times the upper limit of normal or bilirubin levels > 1.5 times the upper limit of normal
5. Severe complications of diabetes mellitus including a history or finding of Stage III or IV diabetic retinopathy (see Appendix B), proteinuria > 2+ by urine dipstick, serum creatinine of >1.8 mg/dl for males or >1.5 mg/dl for females, history of renal transplant, severe peripheral vascular disease, which has resulted in amputation or recent onset of chronic foot ulcers or claudication, or the recent, clinically documented loss a pedal pulse.
6. History of moderate to severe ketoacidosis within the 3 months preceding screening for the study
7. Current drug or alcohol abuse, or a history which in the opinion of the Investigator will impair subject safety or protocol compliance.
8. Current significant cardiovascular, respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and/or hematological disease as evaluated by the Investigator
9. A sexually active woman of childbearing age not actively and consistently practicing birth control by using a medically accepted device or therapy or a woman intending to become pregnant during the study
10. Abnormal ECG, safety lab or physical examination results which, in the opinion of the investigator, render the participation of the subject in the study to be inappropriate or unsafe
11. A history of lack of compliance with medical instructions, recent drug or alcohol abuse, or other reasons which, in the opinion of the investigator, render the participation of the subject in the study to be inappropriate or unsafe

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The frequency of occurrence of hypoglycemia measured quarterly over one year. | 18 months for most subjects

SECONDARY OUTCOMES:
Changes in total daily:Prandial insulin dose, insulin dose, body weight, insulin antibody titers, the effects of insulin antibodies on glycemic control, individual and group mean %HbA1C measured quarterly and over one year. | 18 months for most subjects